CLINICAL TRIAL: NCT03884686
Title: Promote Food. Improving Food-related Quality of Life in Patients With Inflammatory Bowel Disease: a Feasibility Study of a Web-base Educational Intervention.
Brief Title: Promote Food. Improving Food-related Quality of Life in Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAS 241127
Record Dates: First submitted 2018-06-28; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Quality of Life; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: One group will receive intervention and other group will receive usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention (Experimental): Patients allocated to intervention arm will have unlimited free access to a web-based education resource.
  Interventions: Other: Web-based education resource
- Usual care (No Intervention): Patients allocated to usual care will receive all usual care and education opportunities.

INTERVENTIONS:
Other: Web-based education resource — Intervention includes fact sheets, question and answers, short videos featuring patients and/or clinicians.
  Arms: Web-based intervention

SUMMARY:
In previous studies, people with inflammatory bowel disease reported that the disease had a large impact on the psychosocial aspects of eating and drinking, and a high proportion of people felt excluded from social interactions that involved eating and drinking (for example religious, family) and there was considerable uncertainty around how eating will affect bowel function together with feelings of reduced autonomy and high levels of stress and anxiety. These patient experiences may lead to reduced food related quality of life.

This randomised control trial will examine the feasibility of using a web based intervention to improve the food related quality of life of people with inflammatory bowel disease. Fifty eligible participants will be randomised to receive either a 3-month website based intervention or usual care. The feasibility of study design, an estimate of the efficacy of the website intervention and patient experience of the intervention will be assessed after three months.

Patients will be recruited from inflammatory bowel disease outpatient clinics at Guy's and St Thomas' NHS Foundation Trust and Bart's Health NHS Trust in the United Kingdom.

DETAILED DESCRIPTION:
The intervention. The web based intervention has been developed based on the outcomes of a previous study. The website is partially populated with several pages which contain educational material designed for patients newly diagnosed (within the last 12 months) with inflammatory bowel disease. The education material provides information related to different problems, short video clips of patients talking about their problems and ways of managing it, or a patient and health care professional consultation in relation to a particular problem, as well as question and answer fact sheets. In order to make the intervention relevant and acceptable to patients and health care professionals, both these groups were actively involved at each stage of the intervention development. During the 3 month intervention patients will have free and unlimited access to the website. Use of the website during the intervention phase will be monitored by the researcher and weekly emails will be sent to participants who do not engage in the intervention. Monthly emails will be sent to all intervention group patients to encourage engagement with the intervention.

Usual care. The patients randomised to usual care will have access to all usual care, including scheduled appointments and nurse-led telephone helpful. They will not have access to the intervention website.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with either Crohn's disease or ulcerative colitis (collectively called inflammatory bowel disease) within the last 12 months

  * Proof of diagnosis (record of diagnostic endoscopy)
  * Aged 16 years and over
  * People who are experiencing food-related problems as a result of their inflammatory bowel disease (90 points or below, out of possible 145 measured by food related quality of life questionnaire)
  * People consuming a free oral diet
  * Sufficient command of written and spoken English to understand the study documentation and procedures
  * Access to internet and skills and ability to use electronic resources

Exclusion Criteria:

* People diagnosed with inflammatory bowel disease for more than 12 months

  * Diagnosis of indeterminate colitis
  * Hospitalised, nursing home or any other form of institutionalised living
  * Receiving intravenous nutrition, enteral nutrition or oral nutritional support which means that food intake is less than 50% of energy requirements (i.e. their energy from food is less than their energy intake from artificial nutritional support)
  * Diagnoses of other co-morbidities that may have impact on diet e.g. diabetes mellitus, coeliac disease, food allergies (not related to inflammatory bowel disease)
  * Pregnancy or less than 6 months post-partum
  * Inability to give informed consent (due to reduced mental capacity)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-16 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change in food-related quality of life score as measured using validated questionnaire FR-QoL-29 | 3 months
  Measured using validated questionnaire Food-Related Quality of Life (FR-QOL), consisting of 29 questions. Each question is answered on a 5 point Likert scale. The sum of which is the overall score. The minimum score is 29 (low food related quality of life) and maximum 145 (high food related quality of life). A score of less than 90 suggests poor food related quality of life.

SECONDARY OUTCOMES:
Change in United Kingdom inflammatory bowel disease questionnaire score | 3 months
  Measured using validated questionnaire the United Kingdom inflammatory bowel disease questionnaire (UK-IBDQ). This is a global disease specific quality of life questionnaire composed of 32 questions which are scored on a 4 point scale. Minimum score is 32 which indicates very poor quality of life and maximum score is 128 which is optimal quality of life.
Change in disease activity index as measured using validated questionnaires | 3 months
  Measured using validated disease specific questionnaires Harvey Bradshaw Index (HBI) if patient has Crohn's disease. This questionnaire contains five questions. If the patient has ulcerative colitis the simple clinical colitis activity index (SCCAI) questionnaire will be used. It contains six questions. The minimum scores for both questionnaires is 0 and indicates disease is in remission. There are no maximum values but the higher the number the greater severe the disease activity.
Change in presence of anxiety and depression score | 3 months
  Measured using validated questionnaire the hospital anxiety and depression score (HADS). The questionnaire contains 14 questions which are scored from 0 to 4. Seven questions relate to anxiety and seven relate to depression. An anxiety or depression sub-score of 0 suggests absence of anxiety or depression and a sub-score of eight or greater suggests borderline presence of anxiety or depression. A sub-score of 10 or more suggests presence of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Cox SR, Czuber-Dochan W, Wall CL, Clarke H, Drysdale C, Lomer MC, Lindsay JO, Whelan K. Improving Food-Related Quality of Life in Inflammatory Bowel Disease through a Novel Web Resource: A Feasibility Randomised Controlled Trial. Nutrients. 2022 Oct 14;14(20):4292. doi: 10.3390/nu14204292. PMID 36296976